CLINICAL TRIAL: NCT04850248
Title: Scoring Model for Predicting Outcome in Patients With Cardiogenic Shock: From Emergency Room to Intensive Care Unit
Brief Title: Scoring Model for Predicting Outcome in Patients With Cardiogenic Shock
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202103043RIND
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Cardiogenic Shock
Keywords: cardiogenic shock; epidemiography; outcome
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention, this is an observational study — no intervention, this is an observational study

SUMMARY:
This study aims to develop a predictive model for the outcomes of patients with cardiogenic shock

DETAILED DESCRIPTION:
This retrospective observational study will enroll patients with cardiogenic shock admitted to the cardiac care unit. Patient characteristics, clinical events during hospitalization, and laboratory examination findings will be collected and analyzed to determine factors associated with mortality. A nomogram will be developed accordingly and will undergo both internal and external validation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cardiogenic shock
* Admitted to the cardiac care unit (CCU)

Exclusion Criteria:

* Non-cardiogenic shock in origin
* Post open heart surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll patients with who arrived at the emergency department with cardiogenic shock and subsequently admitted to the cardiac care unit.
Sampling Method: Non-Probability Sample
Enrollment: 999 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | through study completion, an average of 1 year
  In-hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Min-Shan Tsai, MD, PhD, Principal Investigator — National Taiwan University Hospital